CLINICAL TRIAL: NCT06303765
Title: Evaluating the Practice Resource for Driving After Stroke (PReDAS): A Concurrent, Multiple Baseline Study
Brief Title: Evaluating the Practice Resource for Driving After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Liliana Alvarez Jaramillo, Assistant Professor, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13Nov2023PReDAS Study
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Stroke, Acute; Driving; Occupational Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: multiple baseline study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PReDAS intervention (Experimental): All participants will receive the PReDAS intervention during the study. As per concurrent multiple baseline designs, each participant will be randomized as to WHEN they receive the PReDAS during the 6 month study period. Baseline lengths will vary from 2 to 5 months.
  Interventions: Other: Practice Resource for Driving After Stroke (PReDAS)

INTERVENTIONS:
Other: Practice Resource for Driving After Stroke (PReDAS) — 1. Provision of written copy of PReDAS for occupational therapist to review
  2. 1:1 online training session to use the PReDAS (1 hour in length)

SUMMARY:
After stroke, individuals must be assessed to determine if they can resume driving. Return to driving is very important to people who have experienced a stroke. Unfortunately, health care providers face challenges in addressing driving after stroke. Common issues include being unsure of the best screening practices, difficulty discussing driving with patients, and challenges making informed recommendations about driving that balance the risk of public safety along with supporting patient goals. Occupational Therapists (OTs) are health care providers that provide screening, assessment, and intervention for driving to individuals who have had a stroke. OTs working in stroke care have highlighted the urgency for evidence-based resources to support practice to address driving with patients. The Practice Resource for Driving After Stroke (PReDAS), is an evidenced-based resource to support the clinical practice of OTs in addressing driving in acute stroke settings. A previous pilot study has demonstrated that the PReDAS is considered useful by both health care providers and patients. Further study is needed to evaluate how the PReDAS can support OTs in addressing driving with patients. The current study proposes to provide the PReDAS as an intervention to OTs working in acute stroke settings to see if the intervention increases OT's self efficacy and clinical reasoning for addressing driving. The study will take repeated measures of self-efficacy and clinical reasoning among participating OTs to determine if the PReDAS intervention supports improved self-efficacy and clinical reasoning.

DETAILED DESCRIPTION:
Background Negotiating return to driving after stroke is a complex process for both clients and health professionals. In many jurisdictions worldwide, there is a mandatory period of driving restriction post-stroke and driving can only be resumed when functional assessments reveal no residual functional impairments that would impact driving ability, including within Canada. Clients experience considerable practical and symbolic challenges when driving status is questioned and community mobility is threatened. Health care providers, including occupational therapists, similarly feel ill-equipped to broach the contentious topic of driving with their clients. As such, extant literature has identified the need for context-specific practice resources for health professionals to navigate the difficult return to driving process with clients following stroke. In response, the Practice Resource for Driving After Stroke (PReDAS) was developed to provide occupational therapists with a comprehensive, stroke-specific, evidence-based resource to inform clinical reasoning for addressing driving in the acute care setting, where initial discussions about driving take place following stroke.

The PReDAS, informed by the Canadian Stroke Best Practice guidelines, includes resources and procedures for 5 key elements including: (1) best practice education for the practitioner, (2) fitness to drive screening, (3), clinical decision-making aids, (4) stakeholder communication and (5) community mobility planning. The PReDAS is not a screening tool, but rather a practice resource for clinicians to address driving post-stroke within the acute care context. The PReDAS aims to guide the practitioner through the process of addressing driving from initial conversations with the client to communicating recommendations. In a recent pilot study, occupational therapists and physicians reported the PReDAS provided a clear and consistent process for addressing driving, enhanced communication and collaboration with the team and patient, and supported clinical decision-making for driving recommendations. Patients similarly agreed the PReDAS was a useful resource to address driving and supported their own decisions surrounding returning to driving. The pilot findings support the need for further evaluation of the PReDAS to support the practice of occupational therapists in addressing driving with clients after stroke.

The goal of the proposed study is to examine the effects of the PReDAS on the clinical reasoning and self-efficacy of occupational therapists to address driving in acute stroke settings. Bandura defines self-efficacy as "beliefs in one's capabilities to organize and execute the courses of action required to produce given attainments". Clinical reasoning is defined as a "complex cognitive process that uses formal and informal thinking strategies to gather and analyze patient information, evaluate the significance of this information and weigh alternative actions".

Methods Design A concurrent multiple-baseline design will be utilized to examine the effects of the PReDAS on clinical reasoning and self-efficacy for addressing driving in acute stroke settings among occupational therapists. While this approach includes a smaller sample size, this design will enable detailed, rich data collection from a smaller, engaged group of participants. Occupational therapists in acute care report driving is important to their practice, but consistently report time constraints in their work, which would likely extend to limited time for research participation as well. As such, a randomized controlled trial design requiring many participants to have sufficient statistical power, would be unrealistic given the characteristics of the target population. Moreover, as constructs such as self-efficacy and clinical reasoning may be dynamic, repeated measures as achieved in a multiple baseline design can demonstrate how constructs change over time.

Participants Eight occupational therapists will be recruited through a variety of methods, including online invitations via social media platforms (Facebook, Twitter), professional networks (Clinical Preceptor Network from Western University, Greater Toronto Area Occupational Therapy Professional Practice Leader Network), and professional associations (Canadian Association of Occupational Therapists and Ontario Society of Occupational Therapists, and Provincial Stroke Networks). Occupational therapists are eligible to participate if they currently practice on an acute stroke unit. To avoid threats to treatment fidelity, occupational therapists are ineligible to participate if there is already a participant enrolled from their local workplace (same physical building), or if they have viewed a copy of the PReDAS previously. Invitations to participate will be shared via social media posts and email. The letter of information and consent from will be provided electronically via QualtricsXM, which will direct prospective participants to provide their email address for communication throughout the study.

PReDAS Intervention To ensure each participant receives the same exposure and training for the PReDAS, each occupational therapist will participate in a 1:1 standardized 1-hour training session. A brief multiple-choice knowledge test will be administered to each participant after the training session to evaluate understanding of the material. Training sessions will occur online via Zoom. Participants will also receive a full-text electronic copy of the PReDAS for use and reference throughout the study.

Instruments Self-efficacy will be measured by the Personal Efficacy and Beliefs Scale (PEBS) which measures self-efficacy regarding work-related skills and tasks. Internal reliability is estimated at .82 from a sample of nurses working in acute care. The validity of the PEBS is supported through positive correlations with similar measures of satisfaction, job performance and organizational commitment. Clinical reasoning will be measured by the Self-Assessment of Clinical Reflection and Reasoning (SACRR) developed to evaluate clinical reasoning among occupational therapists and physiotherapists. Internal consistency has been rated between .87 and .92 as measured by Cronbach's Alpha, and Spearman rank order correlation coefficient for test-retest reliability is rated as "acceptable" at .60.

As the PEBS and SACRR are broad measures of job self-efficacy and clinical reasoning and reflection respectively, the measures were slightly adapted to cue the participants to answer the questions specific to addressing driving in their practice. For example, instead of the following item from the PEBS "I have confidence in my ability to do my job", the item was adapted to "I have confidence in my ability to address driving". As with the PEBS, participants will be cued to answer the SACRR it relates to addressing driving in acute care settings. The adapted PEBS and SACRR surveys are presented in Appendix A and B, respectively.

Demographic data will also be collected including (1) email, (2) first and last name, (3) year of graduation from occupational therapy program, and (4) number of years working in acute stroke settings.

Procedure Design standards for multiple-baseline studies recommend at least three A-B tiers and at least 5 data points. As such, the proposed study will aim to recruit eight occupational therapists and obtain seven data collection points, to accommodate for attrition and exceed minimum standards. Data will be collected for a period of 6 months with data collected at seven points: at baseline, 1,2,3,4, 5 and 6 months. The criterion for introduction of the PReDAS intervention to participants will be determined by number of months from baseline, whereby each participant will be randomly assigned to receive the PReDAS at month 2, 3, 4, or 5, ensuring there is at least one participant in each time frame.

The platform QualtricsXM will be used for consent and data collection. Participants will be emailed an online survey link to review the letter of information and express consent to participate in the study. After indicating consent, participants will be automatically re-directed to a separate demographic survey where participants will generate a unique participant ID. At the required seven data collection timepoints, participants will be contacted via email to complete the PEBS and SACRR and enter their unique participant ID. As the demographic survey that connects the participant's name to their participant ID is separate from the data collection survey, the timing of when each participant received the PReDAS intervention will not be known until data analysis is complete to reduce risk of bias.

Analysis Visual analysis involves systematic procedures to assess patterns and relationships in graphed data from multiple baseline designs. Visual analysis facilitates examination of the efficacy of the intervention across time and subjects and is critical for assessing experimental control. As such, visual analysis will be utilized to evaluate changes in (1) clinical reasoning and self-efficacy both within participants and across participants, and (2) observe the relationship between the introduction of the PReDAS and occupational therapist reported clinical reasoning and self-efficacy.

Tau-U analysis is a widely accepted statistical procedure within single subject designs that: can control for Type I errors, adjust for baseline trend, is less affected by within-case variability, correlates well with other indices (such as visual analysis), and discriminates well at upper and lower limits. Tau-U analyses will be conducted to evaluate the effect size of the PReDAS using the conventions of small (<.20), moderate (.20-0.60), large (0.60-0.80) or very large (>0.80).

Expected Results and Knowledge Mobilization The results of the proposed study will provide further evidence for the use of the PReDAS as a resource to occupational therapists in acute care for addressing driving. This is an important next step to establish the PReDAS as evidence-based resource for occupational therapists in acute stroke settings. Moreover, as the study will employ a multiple baseline design, the findings will not only reveal if the introduction of the PReDAS improves clinical reasoning or self-efficacy but will also permit examination of how these constructs may change over time. A manuscript will be prepared to submit to OTJR: Occupational Therapy Journal of Research to disseminate findings. To reach practicing therapists, a presentation will be submitted to two annual occupational therapy conferences, the Canadian Association of Occupational Therapy (CAOT)] and American Association of Occupational Therapy (AJOT), and a webinar proposal will be submitted to CAOT.

ELIGIBILITY:
Inclusion Criteria:

* Practicing Occupational therapist
* current employment on an acute stroke unit

Exclusion Criteria:

* there is already a participant enrolled who is located on the same stroke unit
* the person already has reviewed a copy of the PReDAS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
clinical reasoning | collected at enrollment and end of month 1,2,3,4,5 and 6
  Measured via the Self-Assessment of Clinical Reasoning and Reflection. Min score=26, max score=130, higher scores= better clinical reasoning
self-efficacy | collected at enrollment and end of month 1,2,3,4,5 and 6
  measured via the Personal Efficacy and Beliefs Scale. min score=10, max=60. higher scores= better self efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Alvarez, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Council of Motor Transport Administrators. (2020). Determining Driver Fitness in Canada: Part 1 A Model for the Administration of Driver Fitness Programs and Part 2: CCMTA Medical Standards for Drivers. https://ccmta.ca/ images/CCMTAMedicalStandardsDec12015finalcleancopyJune20016 edit.bookmarkspdf.pdf
- [Background] Liddle, J., Turpin, M., McKenna, K., Kubus, T., Lambley, S., & McCaffrey, K. (2009). The experiences and needs of people who cease driving after stroke. Brain Impairment, 10(3), 271-281. https://doi.org/10.1375/brim.10.3.271
- [Background] Patomella AH, Johansson K, Tham K. Lived experience of driving ability following stroke. Disabil Rehabil. 2009;31(9):726-33. doi: 10.1080/09638280802306539. PMID 18946806
- [Background] Vander Veen A, Laliberte Rudman D. Rethinking Driving Against Medical Advice: The Situated Nature of Driving After Stroke. Can J Occup Ther. 2022 Dec;89(4):406-416. doi: 10.1177/00084174221114670. Epub 2022 Jul 19. PMID 35854415
- [Background] Korner-Bitensky N, Menon A, von Zweck C, Van Benthem K. Occupational therapists' capacity-building needs related to older driver screening, assessment, and intervention: a Canadawide survey. Am J Occup Ther. 2010 Mar-Apr;64(2):316-24. doi: 10.5014/ajot.64.2.316. PMID 20437919
- [Background] Sangrar, R., Griffith, L. E., Letts, L., & Vrkljan, B. (2018). Examining Occupational Therapists' Awareness of Medical Fitness-to-Drive Legislation Using a Knowledge-to-Action Approach. Topics in Geriatric Rehabilitation, 34(4), 274-282. https://doi.org/10.1097/TGR.0000000000000205
- [Background] Cammarata, M., Mueller, A. S., Harris, J., & Vrkljan, B. (2017). The Role of the Occupational Therapist in Driver Rehabilitation After Stroke. Physical and Occupational Therapy in Geriatrics, 35(1), 20-33. https://doi.org/10.1080/02703181.2016.1277443
- [Background] Vander Veen A, Cammarata M, Renner S, Alvarez L. The Clinical Usefulness of the Practice Resource for Driving after Stroke (PReDAS). Occup Ther Health Care. 2023 Jan;37(1):119-144. doi: 10.1080/07380577.2021.2018751. Epub 2021 Dec 26. PMID 34955088
- [Background] Mountain A, Patrice Lindsay M, Teasell R, Salbach NM, de Jong A, Foley N, Bhogal S, Bains N, Bowes R, Cheung D, Corriveau H, Joseph L, Lesko D, Millar A, Parappilly B, Pikula A, Scarfone D, Rochette A, Taylor T, Vallentin T, Dowlatshahi D, Gubitz G, Casaubon LK, Cameron JI. Canadian Stroke Best Practice Recommendations: Rehabilitation, Recovery, and Community Participation following Stroke. Part Two: Transitions and Community Participation Following Stroke. Int J Stroke. 2020 Oct;15(7):789-806. doi: 10.1177/1747493019897847. Epub 2020 Jan 27. PMID 31983292
- [Background] Bandura, A. (1997). Self efficacy: The exercise of control. Freeman.
- [Background] Simmons B. Clinical reasoning: concept analysis. J Adv Nurs. 2010 May;66(5):1151-8. doi: 10.1111/j.1365-2648.2010.05262.x. Epub 2010 Mar 9. PMID 20337790
- [Background] Ledford, J. R., & Gast, D. L. (2018). Single Case Research Methodology: Applications in Special Education and Behavioural Sciences. Routledge.
- [Background] Murray A, Di Tommaso A, Molineux M, Young A, Power P. Contemporary occupational therapy philosophy and practice in hospital settings. Scand J Occup Ther. 2021 Apr;28(3):213-224. doi: 10.1080/11038128.2020.1750691. Epub 2020 May 1. PMID 32356478
- [Background] Vander Veen A, Holmes J, Tucker P, Alvarez L. Addressing Driving in Acute Care: Perceived Relevance and Competence. Can J Occup Ther. 2024 Mar;91(1):88-99. doi: 10.1177/00084174231182898. Epub 2023 Jun 22. PMID 37350112
- [Background] Riggs, M. L., Warka, J., Babasa, B., Betancourt, R., & Hooker, S. (1994). Development and Validation of Self-Efficacy and Outcome Expectancy Scales for Job-Related Applications. Educational and Psychological Measurement, 54(3), 793-802.
- [Background] O'Brien, K. M., Kearney, M. S., & Sauber, E. (2019). Measuring career and occupational self-efficacy. In M. W. Gallagher & S. J. Lopez (Eds.), Positive psychological assessment: A handbook of models and measures (2nd ed.). (2nd ed., pp. 97-110). American Psychological Association. https://doi.org/10.1037/0000138-007
- [Background] Peterson, J., McGillis Hall, L., O'Brien-Pallas, L., & Cockerill, R. (2011). Job satisfaction and intentions to leave of new nurses. Journal of Research in Nursing, 16(6), 536-548. https://doi.org/10.1177/1744987111422423
- [Background] Royeen, C., Mu, K., Barnett, K., & Luebbeb, A. (2000). Pilot Investigtion: Evaluation of Clinical Refelction and Reasoning. In P. A. H. Crist (Ed.), Innovations in Occupational therapy education (pp. 107-115). American Occupational Therapy Association.
- [Background] Tate. (2018). Multiple-Baseline Designs. In R. Tate & M. Perdices (Eds.), Single-Case Experimental Designs for Clinical Research and Neurorehabilitation Settings (1st ed., pp. 108-130). Routledge. https://doi-org.proxy1.lib.uwo.ca/10.4324/9780429488184
- [Background] Barton, E. E., Lloyd, B. P., Spriggs, A. D., & Gast, D. L. (2018). Visual analysis of graphic data. In J. R. Ledford & D. L. Gast (Eds.), Single Case Research Methodology: Applications in Special Education and Behavioral Sciences (3rd ed., pp. 179-214). https://doi.org/10.4324/9780203521892
- [Background] Fingerhut, J., Xu, X., & Moeyaert, M. (2021). Selecting the proper Tau-U measure for single-case experimental designs: Development and application of a decision flowchart. Evidence-Based Communication Assessment and Intervention, 15(3), 99-114. https://doi.org/10.1080/17489539.2021.1937851
- [Background] Parker RI, Vannest KJ, Davis JL, Sauber SB. Combining nonoverlap and trend for single-case research: Tau-U. Behav Ther. 2011 Jun;42(2):284-99. doi: 10.1016/j.beth.2010.08.006. Epub 2011 Feb 3. PMID 21496513
- [Background] Vannest, K. J., & Ninci, J. (2015). Evaluating intervention effects in single-case research designs. Journal of Counseling and Development, 93(4), 403-411. https://doi.org/10.1002/jcad.12038